CLINICAL TRIAL: NCT07188415
Title: Lower Extremity Gait, Mobility and Balance Confidence in Charcot-Marie-Tooth Patients With Cavovarus Foot Deformity
Brief Title: CMT Gait, Mobility, Balance - AOFAS Grant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bopha Chrea (Other)
Responsible Party: Sponsor-Investigator, Bopha Chrea, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 202503402
Record Dates: First submitted 2025-09-17; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Charcot Marie Tooth Disease (CMT)
Keywords: Gait Biomechanics
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Intervention Model Description: Two groups will be recruited in this study, participants who have a history of surgical correction (OP) and participants who have no history of surgical correction for cavovarus foot deformity but do wear clinically prescribed ankle-foot orthotics (NonOP). Participants will complete valid and reliable tests of physical mobility and balance confidence under the direction and supervision of trained study staff. Individuals in the OP group will complete all activities without an AFO and individuals in the NonOP group will complete activities with and without their clinically prescribed ankle foot orthosis, to determine the effect of AFOs on mobility and balance confidence. NonOP participants will complete all procedures in a randomized order to prevent influence of testing order. Gait kinematics and kinetics will be measured using infra-red motion capture cameras (Vicon Motion Systems Ltd., Denver, CO) and force plates (AMTI, Watertown, MA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- OP (No Intervention): Charcot-Marie-Tooth patients who have undergone surgical correction but do not wear ankle-foot orthoses.
- NonOP (Other): Charcot-Marie-Tooth patients who have not undergone surgical correction, but do wear clinically prescribed ankle-foot orthoses. NonOP subjects will complete study procedures both with and without their AFOs.
  Interventions: Device: Ankle-foot Orthoses

INTERVENTIONS:
Device: Ankle-foot Orthoses — Group 1 will consist of individuals who have CMT and have undergone surgical correction (OP) and Group 2 will be AFO users who have CMT but have not undergone major surgical correction (NonOP).
  Arms: NonOP

SUMMARY:
The overall objective of the proposed research is to begin to better understand the potential benefits and limitations of ankle -foot orthosis (AFO) use in the context of mobility and balance during gait for individuals with Charcot-Marie-Tooth disease (CMT). These benefits will be studied in comparison to those offered by surgical correction. We will accomplish by having subjects undergo mobility and balance tests in our gait analysis lab.

DETAILED DESCRIPTION:
Walking is an important daily activity that is compromised in individuals with neuromuscular conditions. Charcot-Marie-Tooth (CMT) disease is the most common form of inherited peripheral neuropathy, affecting 2.8 million people worldwide and 1 in 2500 in the United States. Amongst patients with CMT, impaired walking is the most significant contributor to reduced quality of life in patients with CMT. Furthermore, these gait deficits result in over 80% of individuals with CMT experiencing a fall or near fall event annually, primarily due to tripping and balance related issues. Ankle foot orthoses (AFOs) are commonly used by individuals with CMT, often with the intent of reducing the risk of falls and restoring a more normal gait pattern. However, AFOs are often bulky, uncomfortable, and can be destabilizing for already weak individuals. Surgical correction offers the advantage of improving limb alignment, reduces bulk, and the arduous nature of donning/doffing a brace. However, surgery is not without risk, potential complications, and post-operative recovery. Scientific evidence to help surgeons determine if an AFO or surgery are optimal for a given patient, especially in the setting of a brace-able foot, remains limited. Recent consensus among expert orthopaedic foot and ankle surgeons agrees that 'There is no evidence-based orthopedic studies to help determine optimal timing for surgery, and there is often contradictory advice from the patient's neurologist, physical therapist, and orthotist regarding the role of an operation. There is a critical need to understand how surgical correction affects mobility, balance confidence, and gait compared to AFO bracing in the native cavovarus foot (non-operatively treated). Without such information, the evidence-based approach to answering this critical question will likely remain unrealized.

ELIGIBILITY:
Inclusion Criteria: 1) Clinical diagnosis and genetic confirmation of CMT, 2) Between the ages of 12 and 75, 3) Able to walk at a slow to moderate pace without an AFO, 3) Able to read and write in English and provide written informed consent. 4) Individuals in the NonOP group must have an AFO prescribed for daily activities. Individuals in the OP group will also have had 5) surgical correction of CMT cavovarus foot deformity focused on muscle balancing and hindfoot correction.

Exclusion Criteria: 1) Other causes or risk factors for peripheral neuropathy (for example diabetes, ETOH abuse), 2) Uncorrected visual impairment, 3) History of musculoskeletal injury requiring surgery 4) loss of plantar protective sensation 5) Pain >4/10 while walking (or an increase in pain during testing of >2/10), 6) Concern by the examiner that the individual will not complete the study. For the NonOP group 7) Previous surgical correction of CMT cavovarus foot deformity focused on muscle balancing and hindfoot correction

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Four-Square Step Test | Baseline
  This test of functional mobility requires rapid stepping and changes in direction, that are often limited by lower limb pathology.
Self-selected Walking Velocity | Baseline
  Participants will be instructed to walk at their "normal comfortable" pace for a 10 m distance. The time traveled between the 2 m mark and 8 m mark is recorded in seconds. Two trials will be completed with 15 seconds rest between trials.
Activity Specific Balance Confidence Scale | Baseline
  The ABC is a well-established survey instrument to assess an individual participant's level of balance confidence during functional activities and takes approximately 3 minutes to complete.
Falls Frequency Questionnaire | Baseline
  Survey asking participants the number of times they fell in the previous 24 hours and the previous week. Participants will also be asked to report the most circumstances most commonly associated with fall events.
Lower Extremity Gait Biomechanics | Baseline
  Measurements include: toe clearance height and ankle dorsiflexion angle during swing, peak ankle plantar flexor moment, and peak ankle push off power.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Medical Campus - North Liberty (MCNL), North Liberty, Iowa, United States

IPD SHARING:
Plan to Share IPD: No